CLINICAL TRIAL: NCT01932372
Title: XELJANZ (REGISTERED) TABLETS 5MG SPECIAL INVESTIGATION (ALL-CASES SURVEILLANCE)
Brief Title: Tofacitinib (Xeljanz) Special Investigation for Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921194
Record Dates: First submitted 2013-07-30; First posted 2013-08-30 (Estimated); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Good Post Marketing Study Practice; Tofacitinib; Xeljanz; Regulatory Post Marketing Commitment Plan
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tofacitinib; Etanercept; Antirheumatic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Tofacitinib (Xeljanz): Tablets 5 mg BID
  Interventions: Drug: Tofacitinib (Xeljanz)
- Standard of Care: Standard of Care for Rheumatoid Arthritis
  Interventions: Drug: Etanercept, other Biologics, Disease-modifying antirheumatic drugs (DMARDs), etc

INTERVENTIONS:
Drug: Tofacitinib (Xeljanz) — 5 mg Tablet BID
  Groups: Tofacitinib (Xeljanz)
Drug: Etanercept, other Biologics, Disease-modifying antirheumatic drugs (DMARDs), etc — Etanercept: 10 to 25 mg twice weekly, or 25 to 50 mg once weekly
  Groups: Standard of Care

SUMMARY:
The objective of this Surveillance is to verify the following subject matters concerning Tofacitinib (Xeljanz) under general practice.

1) Occurrence of adverse reactions, factors that may potentially affect safety and efficacy 2） Long-term safety (particularly, malignant tumors and serious infections) and efficacy

Occurrences of malignant tumors and serious infections will be compared with a control group.

DETAILED DESCRIPTION:
All the patients whom an investigator prescribes the Xeljanz or Standard of Care for rheumatoid arthritis should be registered consecutively until the number of subjects reaches target number in order to extract patients enrolled into the investigation at random.

ELIGIBILITY:
Inclusion Criteria:

* All patients receiving Tofacitinib (Xeljanz)

Exclusion Criteria:

Not Applicable

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with moderately to severely active rheumatoid arthritis who have had an inadequate response or intolerance to over 8 mg Methotrexate for 3 months treatment.
Sampling Method: Probability Sample
Enrollment: 9968 (Actual)
Dates: Start 2013-07-26 (Actual); Primary Completion 2021-08-24 (Actual); Study Completion 2021-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Kuwana M, Sugiyama N, Momohara S, Atsumi T, Takei S, Tamura N, Harigai M, Fujii T, Matsuno H, Takeuchi T, Yamamoto K, Takasaki Y, Tanigawa M, Endo Y, Hirose T, Morishima Y, Yoshii N, Mimori T, Takagi M. Six-month safety and effectiveness of tofacitinib in patients with rheumatoid arthritis in Japan: Interim analysis of post-marketing surveillance. Mod Rheumatol. 2024 Feb 26;34(2):272-286. doi: 10.1093/mr/road063. PMID 37405710
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921194&StudyName=Tofacitinib%20%28Xeljanz%29%20Special%20Investigation%20for%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- XELJANZ (Safety Analysis Set): Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months or 6 months. The dosage can be adjusted as per physician's discretion. Participants who did not meet the eligibility criteria and/or were not assessable for safety were excluded.
- Control (MTX Adherent Comparative Safety Analysis Set): Participants with no experience of treatment with XELJANZ Tablets 5 mg, and received treatment other than XELJANZ Tablets 5 mg for rheumatoid arthritis (RA) were observed for a scheduled period of 36 months. The dosage can be adjusted as per physician's discretion. Participants who did not meet the eligibility criteria and/or were not assessable for safety were excluded.
Period: Overall Study
Arm/Group | XELJANZ (Safety Analysis Set) | Control (MTX Adherent Comparative Safety Analysis Set)
Started (Number of participants for whom CRFs were collected) | 7054 (Number of participants in XELJANZ group for whom CRFs were collected.) | 2598 (Number of participants in Control group for whom CRFs were collected.)
XELJANZ (Safety Analysis Set) (Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months or 6 months. The dosage can be adjusted as per physician's discretion. Participants who did not meet the eligibility criteria and/or were not assessable for safety were excluded.) | 7021 (XELJANZ (Safety analysis set) This is the largest analysis populations in XELJANZ group.) | 2419 (Control (MTX adherent comparative safety analysis set))
XELJANZ (MTX Adherent Safety Analysis Set) (Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months or 6 months. The dosage can be adjusted as per physician's discretion. The MTX adherent safety analysis set was defined as the participants within the safety analysis set who have been poorly controlled even though MTX was used continuously dose of more than 8 mg/week for 3 months or longer.) | 4574 (XELJANZ (MTX adherent safety analysis set) is included in 7021.) | 0
XELJANZ (MTX Adherent Comparative Safety Analysis Set) (Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months. The dosage can be adjusted as per physician's discretion. The MTX adherent comparative safety analysis set was defined as the participants with RA who have been poorly controlled even though MTX was used continuously at a dose of more than 8 mg/week for 3 months or longer, excluding the participants with observation for 6 months or shorter.) | 3731 (XELJANZ (MTX adherent comparative safety analysis set) is included in 7021.) | 0
Completed | 7021 | 2419
Not Completed | 33 | 179
Not completed — Not meeting eligibility criteria | 33 | 179

BASELINE CHARACTERISTICS:
Population: Of the participants who were confirmed completed the study, those who met the eligibility criteria were included in the following analysis sets: XELJANZ safety analysis set, n=7021; Xeljanz MTX adherent safety analysis set, n=4574; Xeljanz MTX adherent comparative safety analysis set, n=3731; and Control MTX adherent comparative safety analysis set, n=2419.
Groups:
- Control (MTX Adherent Comparative Safety Analysis Set): Participants with no experience of treatment with XELJANZ Tablets 5 mg, and received treatment other than XELJANZ Tablets 5 mg for RA were observed for a scheduled period of 36 months. The dosage can be adjusted as per physician's discretion. Participants who did not meet the eligibility criteria and/or were not assessable for safety were excluded.
- Total: Total of all reporting groups
Arm/Group | XELJANZ (Safety Analysis Set) | Control (MTX Adherent Comparative Safety Analysis Set) | Total
Number analyzed (Participants) | 7021 | 2419 | 9440
Age, Customized [Number; unit: Participants] — Population: In the XELJANZ group, safety analysis set corresponds to overall. The MTX adherent safety analysis set is a group of participants who meet the eligibility criteria for MTX among the safety analysis set. The MTX adherent comparative safety analysis set is a group of participants in the safety analysis set who were observed for a scheduled period of 36 months and meet the eligibility criteria for MTX. In the Control group, the MTX adherent comparative safety analysis set corresponds to overall.
  Participants
    <50 years | 1112 | 728 | 1840
    ≥50 and <65 years | 2284 | 905 | 3189
    ≥65 years | 3625 | 786 | 4411
    XELJANZ (MTX adherent safety analysis set) <50 years: number analyzed (Participants) | 4574 | 2419 | 6993
    XELJANZ (MTX adherent safety analysis set) <50 years | 859 | 0 | 859
    XELJANZ (MTX adherent safety analysis set) ≥50 and <65 years: number analyzed (Participants) | 4574 | 2419 | 6993
    XELJANZ (MTX adherent safety analysis set) ≥50 and <65 years | 1632 | 0 | 1632
    XELJANZ (MTX adherent safety analysis set) ≥65 years: number analyzed (Participants) | 4574 | 2419 | 6993
    XELJANZ (MTX adherent safety analysis set) ≥65 years | 2083 | 0 | 2083
    XELJANZ (MTX adherent comparative safety analysis set) <50 years: number analyzed (Participants) | 3731 | 2419 | 6150
    XELJANZ (MTX adherent comparative safety analysis set) <50 years | 705 | 0 | 705
    XELJANZ (MTX adherent comparative safety analysis set) ≥50 and <65 years: number analyzed (Participants) | 3731 | 2419 | 6150
    XELJANZ (MTX adherent comparative safety analysis set) ≥50 and <65 years | 1360 | 0 | 1360
    XELJANZ (MTX adherent comparative safety analysis set) ≥65 years: number analyzed (Participants) | 3731 | 2419 | 6150
    XELJANZ (MTX adherent comparative safety analysis set) ≥65 years | 1666 | 0 | 1666
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In the XELJANZ group, safety analysis set corresponds to overall. The MTX adherent safety analysis set is a group of participants who meet the eligibility criteria for MTX among the safety analysis set. The MTX adherent comparative safety analysis set is a group of participants in the safety analysis set who were observed for a scheduled period of 36 months and meet the eligibility criteria for MTX. In the Control group, the MTX adherent comparative safety analysis set corresponds to overall.
  Participants
    XELJANZ (Safety analysis set) and Control (MTX adherent comparative safety analysis set): Female | 5598 | 1836 | 7434
    XELJANZ (Safety analysis set) and Control (MTX adherent comparative safety analysis set): Male | 1423 | 583 | 2006
    XELJANZ (MTX adherent safety analysis set): number analyzed (Participants) | 4574 | 0 | 4574
    XELJANZ (MTX adherent safety analysis set): Female | 3615 | 0 | 3615
    XELJANZ (MTX adherent safety analysis set): Male | 959 | 0 | 959
    XELJANZ (MTX adherent comparative safety analysis set): number analyzed (Participants) | 3731 | 0 | 3731
    XELJANZ (MTX adherent comparative safety analysis set): Female | 2935 | 0 | 2935
    XELJANZ (MTX adherent comparative safety analysis set): Male | 796 | 0 | 796
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-related Adverse Events or Serious Treatment-related Adverse Events in Participants Who Received XELJANZ
Description: An adverse drug reaction (ADR) was any untoward medical occurrence attributed to XELJANZ in a participant who received XELJANZ. A serious adverse event/adverse drug reaction (SADR) was a treatment-related adverse event resulting in any of the following outcomes or deemed significant for any other reason: death; life-threatening experience (immediate risk of dying); initial or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly. Relatedness to XELJANZ was assessed by the physician.
Time Frame: 36 months
Population: The MTX adherent safety analysis set (n=4574) comprised of participants who received XELJANZ Tablets 5 mg at least once for the treatment of poorly controlled RA despite continuous use of MTX, excluding participants who did not meet the conditions to receive MTX, participated in a clinical trial, or transferred to another hospital.
Measure: Number; unit: Percentage of Participants
Groups:
- XELJANZ (MTX Adherent Safety Analysis Set): Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months or 6 months. The dosage can be adjusted as per physician's discretion. The MTX adherent safety analysis set was defined as the participants within the safety analysis set who have been poorly controlled even though MTX was used continuously at a dose of more than 8 mg/week for 3 months or longer.
Arm/Group | XELJANZ (MTX Adherent Safety Analysis Set)
Number analyzed (Participants) | 4574
Percentage of Participants
  ADR | 41.60
  Serious ADR | 12.88

2. Secondary Outcome: Occurrence of Serious Infection Events
Description: Comparison of time to serious infection between XELJANZ group and control group.
  Hazard ratio (unadjusted): Baseline characteristics are unadjusted Hazard ratio (adjusted 1): Adjusted by propensity score estimated by logistic regression Hazard ratio (adjusted 2): Adjusted by propensity score estimated by random forest Hazard ratio (adjusted 3): Adjusted by propensity score estimated by logistic regression (with upper limit of weighting) Hazard ratio (adjusted 4): Adjusted by propensity score estimated by random forest (with upper limit of weighting)
Time Frame: 12 months
Population: The MTX adherent comparative safety analysis set comprised of participants who satisfied the inclusion criteria and had received XELJANZ Tablets 5 mg or other treatment at least once for the treatment of poorly controlled RA despite continuous use of MTX.
Measure: Number (95% Confidence Interval); unit: Incidence rate; participants /100 PY
Groups:
- XELJANZ (MTX Adherent Comparative Safety Analysis Set): Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months. The dosage can be adjusted as per physician's discretion. The MTX adherent comparative safety analysis set was defined as the participants with RA who have been poorly controlled even though MTX was used continuously at a dose of more than 8 mg/week for 3 months or longer, excluding the participants with observation for 6 months or shorter.
Arm/Group | XELJANZ (MTX Adherent Comparative Safety Analysis Set) | Control (MTX Adherent Comparative Safety Analysis Set)
Number analyzed (Participants) | 3731 | 2419
Incidence rate; participants /100 PY | 6.86 [5.96 to 7.86] | 1.42 [0.97 to 2.00]
Statistical Analysis 1: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Incidence rate ratio (unadjusted) = 4.85, 95% CI 2-sided [3.34 to 7.03]
Statistical Analysis 2: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (unadjusted) = 4.80, 95% CI 2-sided [3.31 to 6.96]
Statistical Analysis 3: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 1) = 2.07, 95% CI 2-sided [0.95 to 4.51]
Statistical Analysis 4: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 2) = 3.81, 95% CI 2-sided [2.24 to 6.47]
Statistical Analysis 5: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 3) = 3.55, 95% CI 2-sided [2.08 to 6.09]
Statistical Analysis 6: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 4) = 3.80, 95% CI 2-sided [2.31 to 6.25]

3. Secondary Outcome: Occurrence of Malignancy
Description: Comparison of time to malignancy between XELJANZ group and control group. The standard incidence ratio (SIR) was calculated using the general Japanese population as the reference population.
  Hazard ratio (unadjusted): Baseline characteristics are unadjusted Hazard ratio (adjusted 1): Adjusted by propensity score estimated by logistic regression Hazard ratio (adjusted 2): Adjusted by propensity score estimated by random forest Hazard ratio (adjusted 3): Adjusted by propensity score estimated by logistic regression (with upper limit of weighting) Hazard ratio (adjusted 4): Adjusted by propensity score estimated by random forest (with upper limit of weighting)
Time Frame: 36 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Incidence rate; participants /100 PY
Arm/Group | XELJANZ (MTX Adherent Comparative Safety Analysis Set) | Control (MTX Adherent Comparative Safety Analysis Set)
Number analyzed (Participants) | 3731 | 2419
Incidence rate; participants /100 PY
  Incidence rate | 1.40 [1.18 to 1.66] | 0.88 [0.66 to 1.15]
  SIR | 1.38 [1.16 to 1.62] | 0.98 [0.73 to 1.28]
Statistical Analysis 1: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Incidence rate ratio (unadjusted) = 1.60, 95% CI 2-sided [1.16 to 2.19]
Statistical Analysis 2: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (unadjusted) = 1.55, 95% CI 2-sided [1.12 to 2.13]
Statistical Analysis 3: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 1) = 1.86, 95% CI 2-sided [1.16 to 2.99]
Statistical Analysis 4: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 2) = 1.61, 95% CI 2-sided [1.06 to 2.43]
Statistical Analysis 5: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 3) = 1.53, 95% CI 2-sided [1.00 to 2.35]
Statistical Analysis 6: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (adjusted 4) = 1.51, 95% CI 2-sided [1.03 to 2.22]

4. Secondary Outcome: Occurrence of Death
Description: Comparison of time to death between XELJANZ group and control group. The standardized mortality ratio (SMR) was calculated using the general Japanese population as the reference population.
  Hazard ratio (unadjusted): Baseline characteristics are unadjusted
Time Frame: 36 months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Mortality rate; participants /100 PY
Arm/Group | XELJANZ (MTX Adherent Comparative Safety Analysis Set) | Control (MTX Adherent Comparative Safety Analysis Set)
Number analyzed (Participants) | 3731 | 2419
Mortality rate; participants /100 PY
  Mortality rate | 0.89 [0.72 to 1.10] | 0.26 [0.15 to 0.43]
  SMR | 1.02 [0.82 to 1.26] | 0.39 [0.23 to 0.64]
Statistical Analysis 1: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Mortality rate ratio (unadjusted) = 3.39, 95% CI 2-sided [1.99 to 5.78]
Statistical Analysis 2: Comparison: XELJANZ (MTX Adherent Comparative Safety Analysis Set) vs Control (MTX Adherent Comparative Safety Analysis Set); Test type: Other; Hazard ratio (unadjusted) = 3.29, 95% CI 2-sided [1.93 to 5.61]

5. Primary Outcome: Change in Disease Activity Based on Simplified Disease Activity Index (SDAI)
Description: The SDAI is the numerical sum of five outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, patient global assessment (PtGA) and physician global assessment (PGA) assessed on 0-10 cm VAS, and C-reactive protein (CRP) (mg/dL). SDAI is defined as follows: ≤3.3, disease remission; >3.3 to ≤11, low disease activity, >11 to ≤26, moderate disease activity; and >26, high disease activity. SDAI was assessed at each evaluation time point and mean change from the start of XELJANZ was calculated with the 95% CI.
Time Frame: Baseline, 1, 6, 12, 24, 36 months
Population: The MTX adherent efficacy analysis set (n=4455) comprised of participants who received XELJANZ Tablets 5 mg at least once for the treatment of poorly controlled RA despite continuous use of MTX, excluding participants who were confirmed ineligible or not assessable for effectiveness. Of the 4455 MTX adherent efficacy analysis set, the participants with available results at each evaluation point are described.
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Groups:
- XELJANZ (MTX Adherent Efficacy Analysis Set) At 1 Month From Baseline; XELJANZ (MTX Adherent Efficacy Analysis Set) At 6 Months From Baseline; XELJANZ (MTX Adherent Efficacy Analysis Set) At 12 Months From Baseline; XELJANZ (MTX Adherent Efficacy Analysis Set) At 24 Months From Baseline; XELJANZ (MTX Adherent Efficacy Analysis Set) At 36 Months From Baseline: Participants who received XELJANZ Tablets 5 mg as indicated in the approved local product document were observed for a scheduled period of 36 months or 6 months. The dosage can be adjusted as per physician's discretion.
Arm/Group | XELJANZ (MTX Adherent Efficacy Analysis Set) At 1 Month From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 6 Months From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 12 Months From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 24 Months From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 36 Months From Baseline
Number analyzed (Participants) | 1937 | 2520 | 1661 | 1227 | 976
Scores on a scale | -10.16 [-10.69 to -9.62] | -14.59 [-15.10 to -14.07] | -15.97 [-16.62 to -15.32] | -16.88 [-17.64 to -16.12] | -17.37 [-18.21 to -16.53]

6. Primary Outcome: Change in Disease Activity Score Based on 28-joints Count (DAS28)
Description: DAS28 is the numerical sum of 4 outcome parameters: tender joint count (TJC) and swollen joint count (SJC) based on a 28-joint assessment, PtGA assessed on 0-10 cm VAS, and the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hour]). DAS28 is defined as follows: <2.6, disease remission; ≥2.6 to <3.2, low disease activity, ≥3.2 to ≤5.1, moderate disease activity; and >5.1, high disease activity. DAS28 was assessed at each evaluation time point and mean change from the start of XELJANZ was calculated with the 95% CI.
Time Frame: Baseline, 1, 6, 12, 24, 36 months
Population: as for outcome 5
Measure: Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | XELJANZ (MTX Adherent Efficacy Analysis Set) At 1 Month From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 6 Months From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 12 Months From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 24 Months From Baseline | XELJANZ (MTX Adherent Efficacy Analysis Set) At 36 Months From Baseline
Number analyzed (Participants) | 1682 | 2119 | 1440 | 1074 | 852
Scores on a scale | -0.98 [-1.04 to -0.92] | -1.52 [-1.58 to -1.46] | -1.67 [-1.75 to -1.59] | -1.82 [-1.91 to -1.73] | -1.86 [-1.96 to -1.76]

ADVERSE EVENTS:
Time Frame: 36 months
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both serious and non-serious events during the study.
Arm/Group | XELJANZ (Safety Analysis Set) | XELJANZ (MTX Adherent Comparative Safety Analysis Set) | Control (MTX Adherent Comparative Safety Analysis Set)
All-Cause Mortality (participants affected / at risk) | 188/7021 | 98/3731 | 16/2419
Serious Adverse Events (participants affected / at risk) | 1351/7021 | 773/3731 | 112/2419
Other Adverse Events (participants affected / at risk) | 1340/7021 | 814/3731 | 28/2419
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | XELJANZ (Safety Analysis Set) (N=7021) | XELJANZ (MTX Adherent Comparative Safety Analysis Set) (N=3731) | Control (MTX Adherent Comparative Safety Analysis Set) (N=2419)
Anaemia (Blood and lymphatic system disorders) | 19 | 9 | 1
Anaemia folate deficiency (Blood and lymphatic system disorders) | 1 | 1 | 0
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 3 | 2 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 7 | 3 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Myelosuppression (Blood and lymphatic system disorders) | 2 | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 2 | 0
Angina pectoris (Cardiac disorders) | 4 | 1 | 1
Angina unstable (Cardiac disorders) | 5 | 3 | 0
Aortic valve stenosis (Cardiac disorders) | 2 | 1 | 0
Arrhythmia (Cardiac disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 11 | 7 | 0
Cardiac failure acute (Cardiac disorders) | 6 | 3 | 0
Cardiac failure chronic (Cardiac disorders) | 2 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 9 | 5 | 1
Cardiac valve disease (Cardiac disorders) | 1 | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 2 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Cataract (Eye disorders) | 4 | 4 | 0
Corneal degeneration (Eye disorders) | 1 | 0 | 0
Corneal perforation (Eye disorders) | 1 | 1 | 0
Eye haemorrhage (Eye disorders) | 1 | 1 | 0
Glaucoma (Eye disorders) | 3 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Anorectal disorder (Gastrointestinal disorders) | 1 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 4 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 2 | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 2 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 5 | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer (Gastrointestinal disorders) | 3 | 2 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 4 | 2 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 1 | 0
Gastric mucosal lesion (Gastrointestinal disorders) | 1 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 8 | 3 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 3 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 3 | 2 | 0
Inguinal hernia (Gastrointestinal disorders) | 3 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 1 | 0
Death (General disorders) | 15 | 9 | 0
Impaired healing (General disorders) | 1 | 1 | 0
Malaise (General disorders) | 2 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Oedema peripheral (General disorders) | 3 | 1 | 0
Perforation (General disorders) | 1 | 1 | 0
Pyrexia (General disorders) | 19 | 11 | 0
Bile duct stone (Hepatobiliary disorders) | 2 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 4 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 2 | 0
Cholecystitis acute (Hepatobiliary disorders) | 5 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 2 | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 9 | 5 | 1
Amyloidosis (Immune system disorders) | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0 | 0
Abscess limb (Infections and infestations) | 3 | 3 | 0
Adenoviral haemorrhagic cystitis (Infections and infestations) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 7 | 6 | 0
Arthritis bacterial (Infections and infestations) | 9 | 8 | 3
Arthritis infective (Infections and infestations) | 3 | 3 | 0
Aspergilloma (Infections and infestations) | 1 | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 1 | 0
Atypical mycobacterial infection (Infections and infestations) | 9 | 7 | 1
Atypical pneumonia (Infections and infestations) | 1 | 1 | 0
Bacteraemia (Infections and infestations) | 4 | 1 | 0
Bacterial infection (Infections and infestations) | 2 | 2 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Bone abscess (Infections and infestations) | 1 | 1 | 1
Bone tuberculosis (Infections and infestations) | 1 | 1 | 0
Bronchiolitis (Infections and infestations) | 1 | 1 | 0
Bronchitis (Infections and infestations) | 18 | 13 | 1
Bronchitis mycoplasmal (Infections and infestations) | 1 | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 5 | 3 | 1
Bursitis infective (Infections and infestations) | 2 | 1 | 0
Cellulitis (Infections and infestations) | 33 | 29 | 2
Cholangitis infective (Infections and infestations) | 1 | 1 | 0
Chronic sinusitis (Infections and infestations) | 1 | 1 | 0
Cystitis (Infections and infestations) | 3 | 1 | 0
Cytomegalovirus chorioretinitis (Infections and infestations) | 2 | 1 | 0
Cytomegalovirus gastroenteritis (Infections and infestations) | 1 | 1 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 1 | 0
Cytomegalovirus viraemia (Infections and infestations) | 1 | 0 | 0
Disseminated varicella zoster virus infection (Infections and infestations) | 7 | 4 | 0
Diverticulitis (Infections and infestations) | 6 | 3 | 1
Endocarditis (Infections and infestations) | 1 | 0 | 0
Enteritis infectious (Infections and infestations) | 5 | 4 | 1
Epididymitis (Infections and infestations) | 1 | 1 | 0
Epiglottitis (Infections and infestations) | 2 | 1 | 0
Escherichia sepsis (Infections and infestations) | 2 | 1 | 0
Extradural abscess (Infections and infestations) | 1 | 1 | 0
Focal peritonitis (Infections and infestations) | 1 | 1 | 0
Fungal infection (Infections and infestations) | 1 | 1 | 0
Fungal sepsis (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 7 | 3 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0 | 0
Hepatitis B reactivation (Infections and infestations) | 3 | 2 | 0
Hepatitis E (Infections and infestations) | 1 | 0 | 0
Herpes dermatitis (Infections and infestations) | 1 | 1 | 0
Herpes ophthalmic (Infections and infestations) | 2 | 0 | 0
Herpes virus infection (Infections and infestations) | 1 | 1 | 0
Herpes zoster (Infections and infestations) | 132 | 82 | 5
Herpes zoster infection neurological (Infections and infestations) | 1 | 1 | 0
Herpes zoster meningitis (Infections and infestations) | 1 | 0 | 0
Herpes zoster meningoencephalitis (Infections and infestations) | 1 | 1 | 0
Herpes zoster oticus (Infections and infestations) | 4 | 2 | 0
Infection (Infections and infestations) | 3 | 1 | 0
Infectious pleural effusion (Infections and infestations) | 6 | 5 | 1
Infective spondylitis (Infections and infestations) | 3 | 2 | 0
Influenza (Infections and infestations) | 11 | 7 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Joint abscess (Infections and infestations) | 1 | 0 | 0
Large intestine infection (Infections and infestations) | 1 | 0 | 0
Liver abscess (Infections and infestations) | 4 | 3 | 0
Localised infection (Infections and infestations) | 2 | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 1 | 0
Mediastinal abscess (Infections and infestations) | 1 | 1 | 0
Medical device site joint infection (Infections and infestations) | 1 | 1 | 0
Meningitis aseptic (Infections and infestations) | 1 | 0 | 0
Meningitis bacterial (Infections and infestations) | 1 | 1 | 0
Muscle abscess (Infections and infestations) | 2 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 2 | 1 | 0
Mycobacterium kansasii infection (Infections and infestations) | 0 | 0 | 1
Mycotic endophthalmitis (Infections and infestations) | 1 | 1 | 0
Necrotising fasciitis (Infections and infestations) | 2 | 2 | 0
Oral herpes (Infections and infestations) | 3 | 2 | 0
Osteomyelitis (Infections and infestations) | 4 | 4 | 0
Otitis media acute (Infections and infestations) | 1 | 1 | 0
Periodontitis (Infections and infestations) | 2 | 1 | 0
Peritonitis (Infections and infestations) | 3 | 1 | 0
Peritonsillitis (Infections and infestations) | 1 | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 32 | 23 | 10
Pneumonia (Infections and infestations) | 140 | 73 | 9
Pneumonia bacterial (Infections and infestations) | 47 | 28 | 4
Pneumonia chlamydial (Infections and infestations) | 2 | 2 | 0
Pneumonia cryptococcal (Infections and infestations) | 2 | 2 | 1
Pneumonia cytomegaloviral (Infections and infestations) | 5 | 4 | 0
Pneumonia herpes viral (Infections and infestations) | 1 | 0 | 0
Pneumonia influenzal (Infections and infestations) | 2 | 2 | 0
Pneumonia klebsiella (Infections and infestations) | 1 | 1 | 0
Pneumonia legionella (Infections and infestations) | 4 | 2 | 0
Pneumonia mycoplasmal (Infections and infestations) | 2 | 1 | 1
Pneumonia pneumococcal (Infections and infestations) | 5 | 2 | 2
Pneumonia pseudomonal (Infections and infestations) | 3 | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 1 | 0
Post procedural infection (Infections and infestations) | 7 | 6 | 0
Pseudomembranous colitis (Infections and infestations) | 3 | 2 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0 | 0
Psoas abscess (Infections and infestations) | 3 | 3 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0 | 0
Purulence (Infections and infestations) | 1 | 0 | 0
Accident (Injury, poisoning and procedural complications) | 2 | 2 | 0
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Atypical femur fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 3 | 2 | 0
Comminuted fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Compression fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 3 | 3 | 0
Dislocation of vertebra (Injury, poisoning and procedural complications) | 2 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 64 | 35 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 31 | 17 | 0
Femur fracture (Injury, poisoning and procedural complications) | 22 | 15 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 4 | 3 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foreign body in gastrointestinal tract (Injury, poisoning and procedural complications) | 2 | 2 | 0
Fracture (Injury, poisoning and procedural complications) | 4 | 2 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 3 | 2 | 0
Heat illness (Injury, poisoning and procedural complications) | 2 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 11 | 6 | 0
Ilium fracture (Injury, poisoning and procedural complications) | 2 | 1 | 0
Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 3 | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 3 | 0 | 0
Meniscus injury (Injury, poisoning and procedural complications) | 2 | 1 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0
Near drowning (Injury, poisoning and procedural complications) | 1 | 1 | 0
Open fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 8 | 6 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 0
Blood pressure decreased (Investigations) | 2 | 1 | 0
C-reactive protein increased (Investigations) | 3 | 2 | 0
CSF volume decreased (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 3 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 9 | 3 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Ankle deformity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 7 | 5 | 0
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Atlantoaxial subluxation (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 4 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Finger deformity (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 6 | 4 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Joint destruction (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 10 | 3 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 7 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 5 | 4 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 0
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Anal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 7 | 4
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Castleman's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Cervix carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Chondromatosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 30 | 21 | 3
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 4 | 3
Epstein-Barr virus associated lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3 | 0
External ear neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Extranodal marginal zone B-cell lymphoma (MALT type) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Gastric adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 15 | 3
Gastric cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 1
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Leser-Trelat sign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 5 | 1
Lung carcinoma cell type unspecified stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 22 | 11 | 5
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 6 | 2
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 8 | 4
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 0
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Altered state of consciousness (Nervous system disorders) | 1 | 0 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 1 | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 2 | 2 | 1
Brain stem infarction (Nervous system disorders) | 1 | 1 | 0
Carotid artery aneurysm (Nervous system disorders) | 1 | 1 | 0
Cerebellar haemorrhage (Nervous system disorders) | 3 | 1 | 0
Cerebellar infarction (Nervous system disorders) | 2 | 1 | 0
Cerebral artery embolism (Nervous system disorders) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 8 | 7 | 0
Cerebral infarction (Nervous system disorders) | 12 | 8 | 1
Cubital tunnel syndrome (Nervous system disorders) | 1 | 1 | 0
Dementia (Nervous system disorders) | 4 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 4 | 3 | 0
Facial paralysis (Nervous system disorders) | 2 | 1 | 0
Frontotemporal dementia (Nervous system disorders) | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Intracranial aneurysm (Nervous system disorders) | 2 | 1 | 0
Lacunar infarction (Nervous system disorders) | 3 | 2 | 0
Loss of consciousness (Nervous system disorders) | 2 | 1 | 0
Mononeuropathy multiplex (Nervous system disorders) | 1 | 0 | 0
Monoplegia (Nervous system disorders) | 2 | 2 | 0
Myelopathy (Nervous system disorders) | 4 | 2 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0
Normal pressure hydrocephalus (Nervous system disorders) | 2 | 2 | 0
Phrenic nerve paralysis (Nervous system disorders) | 1 | 0 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 1 | 0
Device connection issue (Product Issues) | 1 | 1 | 0
Device loosening (Product Issues) | 2 | 2 | 0
Completed suicide (Psychiatric disorders) | 3 | 2 | 0
Depression (Psychiatric disorders) | 3 | 2 | 0
Depressive symptom (Psychiatric disorders) | 1 | 1 | 0
Eating disorder (Psychiatric disorders) | 1 | 1 | 0
Schizophrenia (Psychiatric disorders) | 2 | 2 | 0
Acute kidney injury (Renal and urinary disorders) | 6 | 4 | 0
Bladder disorder (Renal and urinary disorders) | 1 | 1 | 0
Calculus urethral (Renal and urinary disorders) | 1 | 0 | 0
Calculus urinary (Renal and urinary disorders) | 2 | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 5 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 1 | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 1 | 0
End stage renal disease (Renal and urinary disorders) | 1 | 0 | 0
Glomerulonephritis membranous (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 2 | 1 | 0
Henoch-Schonlein purpura nephritis (Renal and urinary disorders) | 1 | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 1 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 2 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 0 | 1
Pelvic haemorrhage (Reproductive system and breast disorders) | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 6 | 3 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Diffuse panbronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 83 | 39 | 6
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 5 | 4 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 12 | 4 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pemphigus (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Cataract operation (Surgical and medical procedures) | 2 | 0 | 0
Foot operation (Surgical and medical procedures) | 1 | 0 | 0
Gastrectomy (Surgical and medical procedures) | 1 | 1 | 0
Hip arthroplasty (Surgical and medical procedures) | 1 | 1 | 0
Hospitalisation (Surgical and medical procedures) | 1 | 0 | 0
Intra-thoracic aortic aneurysm repair (Surgical and medical procedures) | 1 | 1 | 0
Joint arthroplasty (Surgical and medical procedures) | 2 | 2 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 2 | 2 | 0
Aortic aneurysm rupture (Vascular disorders) | 2 | 1 | 1
Aortic dissection (Vascular disorders) | 9 | 3 | 0
Artery dissection (Vascular disorders) | 1 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 10 | 7 | 1
Embolism venous (Vascular disorders) | 1 | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 1 | 0
Peripheral artery occlusion (Vascular disorders) | 1 | 1 | 0
Peripheral embolism (Vascular disorders) | 1 | 1 | 0
Rheumatoid vasculitis (Vascular disorders) | 4 | 3 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 8 | 4 | 2
Splenomegaly (Blood and lymphatic system disorders) | 1 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 7 | 2 | 0
Myocardial rupture (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 1 | 0
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0 | 0
Macular fibrosis (Eye disorders) | 1 | 1 | 0
Necrotising retinitis (Eye disorders) | 1 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 0
Diabetes insipidus (Endocrine disorders) | 1 | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1 | 0
Scleritis (Eye disorders) | 1 | 0 | 0
Uveitis (Eye disorders) | 2 | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 4 | 2 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 1 | 0
Mechanical ileus (Gastrointestinal disorders) | 2 | 0 | 0
Melaena (Gastrointestinal disorders) | 3 | 2 | 0
Mesenteric panniculitis (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic disorder (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatic mass (Gastrointestinal disorders) | 2 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 4 | 2 | 0
Peptic ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Retroperitoneal fibrosis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 2 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 3 | 0
Sudden death (General disorders) | 4 | 3 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Liver disorder (Hepatobiliary disorders) | 4 | 2 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0 | 0
Immune reconstitution inflammatory syndrome (Immune system disorders) | 1 | 1 | 0
Pyelonephritis (Infections and infestations) | 23 | 12 | 3
Pyelonephritis acute (Infections and infestations) | 6 | 4 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Salpingitis (Infections and infestations) | 1 | 1 | 0
Sepsis (Infections and infestations) | 25 | 16 | 1
Septic shock (Infections and infestations) | 7 | 3 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0
Sinusitis fungal (Infections and infestations) | 1 | 1 | 0
Skin infection (Infections and infestations) | 1 | 0 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 0 | 0
Systemic mycosis (Infections and infestations) | 1 | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 1 | 0
Tonsillitis bacterial (Infections and infestations) | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 31 | 14 | 0
Varicella (Infections and infestations) | 3 | 3 | 0
Varicella zoster pneumonia (Infections and infestations) | 2 | 1 | 0
Varicella zoster virus infection (Infections and infestations) | 1 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 12 | 6 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pneumoconiosis (Injury, poisoning and procedural complications) | 1 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 3 | 3 | 0
Silicosis (Injury, poisoning and procedural complications) | 1 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 37 | 18 | 0
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0 | 0
Suture rupture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 16 | 11 | 1
Thermal burn (Injury, poisoning and procedural complications) | 1 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 5 | 4 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 4 | 2 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 4 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Influenza virus test positive (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 13 | 7 | 0
Neutrophil count decreased (Investigations) | 2 | 1 | 0
Platelet count decreased (Investigations) | 5 | 2 | 0
Protein urine present (Investigations) | 2 | 0 | 0
Urinary occult blood positive (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 2 | 0
Marasmus (Metabolism and nutrition disorders) | 1 | 1 | 0
Polychondritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Polymyositis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 3 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 48 | 26 | 0
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Wrist deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Metastases to pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 5 | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 6 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Pharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2 | 0
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 3 | 3
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Sarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 5 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 4 | 2 | 0
Putamen haemorrhage (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 2 | 1 | 0
Spinal subarachnoid haemorrhage (Nervous system disorders) | 1 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 6 | 2 | 1
Thalamus haemorrhage (Nervous system disorders) | 3 | 3 | 0
Thrombotic cerebral infarction (Nervous system disorders) | 1 | 0 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 2 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 1 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0 | 0
Ureterolithiasis (Renal and urinary disorders) | 2 | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rheumatoid lung (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Status asthmaticus (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 10 | 5 | 0
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Ostectomy (Surgical and medical procedures) | 1 | 1 | 0
Oxygen therapy (Surgical and medical procedures) | 1 | 1 | 0
Rotator cuff repair (Surgical and medical procedures) | 1 | 1 | 0
Synovectomy (Surgical and medical procedures) | 1 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 1 | 0
Varicose vein (Vascular disorders) | 2 | 2 | 0
Vasculitis (Vascular disorders) | 3 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | XELJANZ (Safety Analysis Set) (N=7021) | XELJANZ (MTX Adherent Comparative Safety Analysis Set) (N=3731) | Control (MTX Adherent Comparative Safety Analysis Set) (N=2419)
Hepatic function abnormal (Hepatobiliary disorders) | 284 | 194 | 3
Bronchitis (Infections and infestations) | 167 | 98 | 2
Herpes zoster (Infections and infestations) | 547 | 325 | 15
Nasopharyngitis (Infections and infestations) | 203 | 124 | 1
Lymphocyte count decreased (Investigations) | 170 | 95 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 214 | 124 | 7

LIMITATIONS AND CAVEATS:
According to the protocol, only three events, Serious Infection, Malignancy, and Death were collected in the control group for comparison with the Xeljanz group and other serious AEs or non-serious AEs were not to be collected although all AEs were collected in Xeljanz group. However several serious and non-serious AEs other than three events were incidentally reported by the investigators in the control group. Note that these AEs do not represent all AEs occurred in the control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/72/NCT01932372/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/72/NCT01932372/SAP_001.pdf